CLINICAL TRIAL: NCT04753905
Title: Surgical Guide for Thoracic Pedicle Screw Instrumentation in Scoliosis Correction Surgery
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: V110C-099
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Surgical Guide for Thoracic Pedicle Screw Instrumentation in Scoliosis Correction Surgery

ELIGIBILITY:
Inclusion Criteria:

* Scoliosis patients

Exclusion Criteria:

* None

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with scoliosis and the cobb angle exceeds over 50 degree.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The accuracy of surgical guile | 1 year
  To evaluate the accuracy of surgical guide, we use the image during surgery to determine whether it's accurate.

CONTACTS AND LOCATIONS:
Locations (1):
- Teipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No